CLINICAL TRIAL: NCT03214432
Title: Return to Work After Mild Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: Rigshospitalet, Denmark (Other); Sygekassernes Helsefond (Other)
Responsible Party: Principal Investigator, Heidi Jeannet Graff, Ph.d. student, University of Copenhagen
Other Study IDs: mTBI-HJG-2017
Record Dates: First submitted 2017-07-05; First posted 2017-07-11 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Mild Traumatic Brain Injury; Concussion, Mild
Keywords: Mild traumatic brain injury; Concussion; Labour market affiliation; Return to work; Sickness absence; Long-term sickness absence; Disability pension
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- mild traumatic brain injury cohort: Patients with mild traumatic brain injury were defined as hospital admitted, emergency or outpatient treated, who were assigned the ICD-10 code for concussion (ICD-10 S06.0) in the national patient register at hospital discharge from the 1st of January 2003 - 31st of December 2007. Patients were working age adults between 18-60 years old and gainfully occupied or deemed available for work the week before the injury.
- non-injured control group: Controls were randomly selected from the Population register who were between 18-60 years old, had no diagnosis of mild traumatic brain injury during the period 1st of January 2003 - 31st of December 2007 and were gainfully occupied or deemed available for work the week preceding the time of injury. One control was matched for each mTBI case on gender, municipality and age (year of birth +/- 0,5 years). In case of no matching control the age criterion was expanded to (year of birth +/- 1 year), if still no matching control the age criterion was further expanded to (year of birth +/- 2 year). Additionally, controls were excluded according to the same criteria as the included cases.

SUMMARY:
Background:

Patients with mild traumatic brain injury can to some extend experience long-term physical, cognitive, social and behavioral deficits, which have serious implications for employment trajectories and financial independence. These deficits have shown to be more pronounced in women. High socio-economic position such as income, level of education and employment status before the accident have shown to affect return to work. But also cohabitation status, ethnicity and health are important factors. Previously studies are typically self-report studies, and are often small and may suffer from selection bias due to patient nonresponse.

Aim:

The aim of this study is to describe no return to work among patients with mild traumatic brain injury in Denmark and to examine how factors such as age, gender, cohabitation status, socio-economic and pre-injury health factors affect no return to work up to 5 years post-injury.

Hypothesis:

We hypothesize that most patients with mild traumatic brain injury return to work within work 6 months post-injury, and that patients with mild traumatic brain injury injury receive more social transfer payments compared to the general population.

Additionally, we hypothesize that low socio economic position, comorbidities and being single are associated with prolonged no return to work.

Methods:

The present study is an observational national register-based cohort study with long-term follow up of patients with mild traumatic brain injury from 1st of January 2008 - 31st of December 2012 in Denmark. Patients aged 18-60 years diagnosed with concussion from 1st of January 2003-31st of December 2007 in the national patient register will be included in the study. Data will be retrieved from several national databases, including the DREAM database containing data on social benefits and reimbursements.

Primary outcome is no-return to work (nRTW) due to any cause and the following four secondary outcomes are graded and should be regarded as a continuum ranging from health related nRTW, limited nRTW, permanently nRTW and mortality.

The results will be published as two separate scientific articles.

ELIGIBILITY:
Inclusion Criteria:

* ICD-10 code for concussion as action diagnosis (ICD-10: S06.0)
* Working age adults between 18-60 years old at the time of injury
* Gainfully occupied or deemed available for work the week preceding the time of injury

Exclusion Criteria:

* Patients were excluded if they were hospital treated and diagnosed with other major neurological injuries such as spinal cord and column injuries and traumatic brain injuries (TBI) besides the concussion at baseline.
* Patients were excluded, who 5 years prior to baseline (1st of January 1998 - 31st of December 2002) had sustained major neurological impairments including concussions.
* Patients outside of the age limit
* Patients not resident in Denmark
* Patients on unemployment benefits and not economically active at the time of injury

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with mild traumatic brain injury were hospital admitted, emergency or outpatient treated and identified on the basis of ICD-10 codes in the National Patient Register from the 1st of January 2003 - 31st of December 2007.
  Patients were included if they were registered in the national patient register database with concussion (ICD-10 S06.0) as primary diagnosis.
Sampling Method: Probability Sample
Enrollment: 38372 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-07-04 (Actual)

PRIMARY OUTCOMES:
nRTW | 5 years follow up
  No-return to work up to 5 years post-injury. nRTW is defined as receiving social transfer payments in any given week during the follow-up period. If no social benefit is given in the DREAM register, it is assumed the patient is gainfully occupied or self-supporting.

SECONDARY OUTCOMES:
Health related nRTW | 5 years follow up
  Health related nRTW is defined as a combined effect of social transfer payments given in case of short or long-term sickness absence. If social transfer payments are granted due to illness it is assumed that the patient is not gainfully working or job seeking.
Limited nRTW | 5 years follow up
  Limited nRTW is defined as a joint effect of several outcome measures granted citizens with permanent reduced work capacity. If no social transfer payments are given, it is assumed that the patients are gainfully occupied or self-supporting.
Permanently nRTW | 5 years follow up
  Individuals between 18-60 years who have permanently reduced work capacity and unable to return to work after injury can be granted disability pension (DP) after an extensive municipal assessment. DP would only be granted persons who have no work capacity left. This outcome includes disability pension and mortality and is regarded as a permanent exit from the labour market.
Mortality | 5 years follow up
  Data on mortality was retrieved from the DREAM register and the proportion of mortality will be assessed during the 5 year follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Hana M Rytter, Study Director — Department of Psychology
Locations (1):
- Department of Psychology, University of Copenhagen, Copenhagen, Copenhagen K, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Graff HJ, Siersma V, Moller A, Kragstrup J, Andersen LL, Egerod I, Mala Rytter H. Premorbid risk factors influencing labour market attachment after mild traumatic brain injury: a national register study with long-term follow-up. BMJ Open. 2019 Apr 11;9(4):e027297. doi: 10.1136/bmjopen-2018-027297. PMID 30975684
- [Derived] Graff HJ, Siersma V, Moller A, Kragstrup J, Andersen LL, Egerod I, Mala Rytter H. Labour market attachment after mild traumatic brain injury: nationwide cohort study with 5-year register follow-up in Denmark. BMJ Open. 2019 Apr 11;9(4):e026104. doi: 10.1136/bmjopen-2018-026104. PMID 30975680